CLINICAL TRIAL: NCT02572362
Title: Estimation of Second Cancer Risk in Patients Planned With Different Radiotherapy Regimes for Rectal Cancer - A Planning Study and Model-based Analysis
Brief Title: Secondary Cancer Risk After Radiation Therapy for Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Kantonsspital Graubuenden (Other)
Collaborators: Klinik Hirslanden, Zurich (Other)
Responsible Party: Principal Investigator, Daniel Rudolf Zwahlen, MD, MBA, Kantonsspital Graubuenden
Other Study IDs: KEK-ZH-Nr. 2014-0255
Record Dates: First submitted 2015-10-04; First posted 2015-10-08 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Neoplasms, Second Primary
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention in this retrospective study — No Intervention in this retrospective Analysis. All patients included did receive Radiation therapy Independent of this study

SUMMARY:
Retrospective study comparing dose distribution of 3D conformal radiotherapy (3DCRT) and volumetric-modulated arc therapy (VMAT) to estimate secondary cancer risk for patients having had radiation therapy for rectal cancer. Twenty-five patients are included in this study. Planning CT scans are used for comparison of dose distribution and calculation of second cancer risk.

DETAILED DESCRIPTION:
A model-based Analysis calculating the organ-specific excess lifetime attributable risk using the planning CT data sets of 25 patients to estimate second cancer risk for patients after radiotherapy for rectal cancer comparing conventional 3DCRT with VAMT techniques.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female > 18 years of age
* pre or postoperative radiation therapy for rectal cancer
* Planning CT

Exclusion Criteria:

* Planning CT not available

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having had radiation therapy for rectal cancer. Estimation of second cancer risk using data from planning CTs comparing dose Distribution using different Radiation therapy techniques (3DCRT vs VMAT).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Calculation of the organ-specific excess lifetime attributable risk (LAR) (%) | 60 years (model-based calculation)
  LAR is calculated for variable Ages at exposure

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Zwahlen, MD, MBA, Principal Investigator — Kantonsspital Graubuenden
Locations (1):
- Klinik Hirslanden, Institute for Radiotherapy, Zurich, Switzerland

REFERENCES:
- [Derived] Zwahlen DR, Bischoff LI, Gruber G, Sumila M, Schneider U. Estimation of second cancer risk after radiotherapy for rectal cancer: comparison of 3D conformal radiotherapy and volumetric modulated arc therapy using different high dose fractionation schemes. Radiat Oncol. 2016 Nov 10;11(1):149. doi: 10.1186/s13014-016-0723-6. PMID 27832799